CLINICAL TRIAL: NCT04409262
Title: A Phase III, Randomized, Double-Blind, Multicenter Study to Evaluate the Efficacy and Safety of Remdesivir Plus Tocilizumab Compared With Remdesivir Plus Placebo in Hospitalized Patients With Severe COVID-19 Pneumonia
Brief Title: A Study to Evaluate the Efficacy and Safety of Remdesivir Plus Tocilizumab Compared With Remdesivir Plus Placebo in Hospitalized Participants With Severe COVID-19 Pneumonia
Acronym: REMDACTA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA42511; 2020-002275-34 (EudraCT Number)
Record Dates: First submitted 2020-05-28; First posted 2020-06-01 (Actual); Results first posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — remdesivir; tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Remdesivir + Tocilizumab (RDV+TCZ) (Experimental): Participants assigned to the RDV+TCZ arm will receive a 10-day treatment course of RDV, plus one infusion of TCZ on Day 1.
  Interventions: Drug: Remdesivir; Drug: Tocilizumab
- Remdesivir + Placebo (RDV+Placebo) (Active Comparator): Participants assigned to the RDV+ placebo arm will receive a 10-day treatment course of RDV, plus one infusion of TCZ-placebo on Day 1.
  Interventions: Drug: Remdesivir; Drug: Placebo

INTERVENTIONS:
Drug: Remdesivir — Participants will receive intravenous (IV) RDV
Drug: Tocilizumab — Participants will receive IV TCZ
  Arms: Remdesivir + Tocilizumab (RDV+TCZ)
Drug: Placebo — Participants will receive IV placebo matched to TCZ
  Arms: Remdesivir + Placebo (RDV+Placebo)

SUMMARY:
This study will evaluate the efficacy and safety of combination therapy with remdesivir plus tocilizumab compared with remdesivir plus placebo in hospitalized patients with COVID-19 pneumonia.

ELIGIBILITY:
Inclusion Criteria

* Hospitalized with COVID-19 pneumonia confirmed per a positive polymerase chain reaction (PCR) of any specimen (e.g., respiratory, blood, urine, stool, other bodily fluid) and evidenced by chest X-ray or CT scan
* Requiring more than 6 L/min supplemental oxygen to maintain SpO2 > 93%
* Agrees to not participate in another clinical trial for the treatment of COVID-19 while participating in this study

Exclusion Criteria

* Known severe allergic reactions to tocilizumab or other monoclonal antibodies
* Known hypersensitivity to remdesivir, the metabolites, or formulation excipients
* Active tuberculosis (TB) infection
* Suspected active bacterial, fungal, viral, or other infection (besides COVID-19)
* In the opinion of the investigator, progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatments
* Treatment with immunosuppressive or immunomodulatory therapy (including tocilizumab) within the past 3 months
* Concurrent treatment with other agents with actual or possible direct-acting antiviral activity against SARS-CoV-2 within 24 hours prior to study drug dosing. In addition, participants with prior or current treatment with > 2 doses of remdesivir for COVID-19 are excluded
* Participating in other drug clinical trials
* Estimated glomerular filtration rate (eGFR) < 30 mL/min (including patients receiving hemodialysis or hemofiltration)
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 x upper limit of normal (ULN) detected within 24 hours of screening (according to local laboratory reference ranges)
* Absolute neutrophil count (ANC) < 1000/uL at screening
* Platelet count < 50,000/uL at screening
* Body weight < 40 kg
* Treatment with an investigational drug within 5 half-lives or 30 days (whichever is longer) of randomization

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 649 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (54):
- United States (38):
  - Valleywise Health Medical Center, Phoenix, Arizona
  - eStudySite - Chula Vista - PPDS, Chula Vista, California
  - Hoag Hospital Irvine, Irvine, California
  - Providence St Johns Health Center, Santa Monica, California
  - Yale University School of Medicine; HIV Clinical Trials Program, New Haven, Connecticut
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Holy Cross Hospital Inc, Fort Lauderdale, Florida
  - Larkin Community Hospital Palm Springs Campus (Hialeah), Hialeah, Florida
  - University of Miami Miller School of Medicine; Clinical Reseach Building, Miami, Florida
  - Larkin Community Hospital, South Miami, Florida
  - St Luke's Health System; Rheumatology Research, Boise, Idaho
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Henry Ford Medical Center, Novi, Michigan
  - St. Michael'S Medical Center, Newark, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - Wyckoff Heights Medical Center, Staten Island, New York
  - Novant Health Clinical Research, Charlotte, North Carolina
  - OhioHealth Research Institute, Columbus, Ohio
  - Providence Saint Vincent's Medical Center, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - The Liver Institute at Methodist Dallas, Arlington, Texas
  - Baylor Scott and White Medical Center - College Station, College Station, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Ben Taub General Hospital - HCHD, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Baylor Scott & White Medical Center - Irving, Irving, Texas
  - Baylor Scott & White Hospital - Plano, Plano, Texas
  - Baylor Scott & White Health, Temple, Texas
  - Intermountain LDS Hospital, Salt Lake City, Utah
  - The Providence Regional Medical Center Everett, Everett, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
- Brazil (7):
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Hospital Nossa Senhora das Graças; Setor de Pesquisa em Neurologia, Curitiba, Paraná
  - Instituto de Pesquisa Clinica Evandro Chagas - IPEC FIOCRUZ, Rio de Janeiro, Rio de Janeiro
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Instituto de Infectologia Emilio Ribas, São Paulo, São Paulo
  - Instituto do Coração - HCFMUSP, São Paulo, São Paulo
- Russia (4):
  - Medsi Clinic, Moscow, Adygeya Republic
  - O.M. Filatov City Clinical Hospital #15; Department of Surgery, Moskva, Moscow Oblast
  - City Pokrovskaya Hospital, Saint Petersburg, Sankt-Peterburg
  - City Clinical Hospital # 52, Moscow
- Spain (5):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Principe de Asturias; Medicina Interna - Servicio de Enfermedades Infecciosas, Alcalá de Henares, Madrid
  - Hospital Universitario HM Torrelodones, Torrelodones, Madrid
  - Hospital General Universitario de Guadalajara, Guadalajara
  - Hospital Universitario Fundacion Jimenez Diaz., Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with severe COVID-19 pneumonia
Groups:
- Remdesivir + Placebo (RDV+PBO): Participants were to receive a 200 mg intravenous (IV) loading dose of RDV, followed by one infusion of PBO on Day 1. Participants were then to be given a 100 mg once daily IV maintenance dose of RDV from Days 2-10, with discontinuation at discharge whether or not 10 days of RDV dosing were completed. One additional infusion of PBO was allowed 8-24 hours after the first for participants with sustained fever or clinically significant worsening of signs or symptoms.
- Remdesivir + Tocilizumab (RDV+TCZ): Participants were to receive a 200 mg intravenous (IV) loading dose of RDV, followed by one infusion of TCZ on Day 1. Participants were then to be given a 100 mg once daily IV maintenance dose of RDV from Days 2-10, with discontinuation at discharge whether or not 10 days of RDV dosing were completed. One additional infusion of TCZ was allowed 8-24 hours after the first for participants with sustained fever or clinically significant worsening of signs or symptoms.
Period: Overall Study
Arm/Group | Remdesivir + Placebo (RDV+PBO) | Remdesivir + Tocilizumab (RDV+TCZ)
Started | 215 | 434
Completed | 140 | 300
Not Completed | 75 | 134
Not completed — Adverse Event | 0 | 2
Not completed — Death | 55 | 97
Not completed — Lost to Follow-up | 12 | 23
Not completed — Lack of Staff | 0 | 1
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 5 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remdesivir + Placebo (RDV+PBO) | Remdesivir + Tocilizumab (RDV+TCZ) | Total
Number analyzed (Participants) | 215 | 434 | 649
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.2 (13.6) | 60.1 (13.3) | 59.5 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 167 | 240
  Male | 142 | 267 | 409
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 125 | 209 | 334
  Not Hispanic or Latino | 88 | 208 | 296
  Unknown or Not Reported | 2 | 17 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 4 | 8
  Asian | 5 | 17 | 22
  Native Hawaiian or Other Pacific Islander | 3 | 7 | 10
  Black or African American | 20 | 52 | 72
  White | 154 | 282 | 436
  More than one race | 2 | 9 | 11
  Unknown or Not Reported | 27 | 63 | 90

OUTCOME MEASURES:

1. Primary Outcome: Time to Hospital Discharge or "Ready for Discharge" up to Day 28
Description: Defined as days from randomization to hospital discharge or "Ready for Discharge" not followed by ordinal scale category >1, hospital readmission or death. Hospital discharge or "Ready for Discharge" is defined as an ordinal score of 1 on the 7-point ordinal scale. Participants who die are censored at Day 28.
  1. Discharged (or "ready for discharge" as evidenced by normal temperature and respiratory rate, and stable oxygen saturation on ambient air or </= 2L supplemental oxygen)
  2. Non-intensive care unit (ICU) hospital ward (or "ready for hospital ward") not requiring supplemental oxygen
  3. Non-ICU hospital ward (or "ready for hospital ward") requiring supplemental oxygen
  4. ICU or non-ICU hospital ward, requiring non-invasive ventilation or high-flow oxygen
  5. ICU, requiring intubation and mechanical ventilation
  6. ICU, requiring extracorporeal membrane oxygenation (ECMO) or mechanical ventilation and additional organ support (e.g., vasopressors, renal replacement therapy)
  7. Death
Time Frame: Up to Day 28
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Remdesivir + Placebo (RDV+Placebo) - mITT Population; Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population: The mITT population included all randomized participants who received any amount of TCZ or placebo (PBO), with participants grouped according to treatment assigned at randomization.
Arm/Group | Remdesivir + Placebo (RDV+Placebo) - mITT Population | Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population
Number analyzed (Participants) | 210 | 430
days | 14.0 [11.0 to 16.0] | 14.0 [12.0 to 15.0]
Statistical Analysis 1: Comparison: Remdesivir + Placebo (RDV+Placebo) - mITT Population vs Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population; Test type: Superiority; p = 0.7414, Log Rank; Hazard Ratio (HR) = 0.965, 95% CI 2-sided [0.78 to 1.19]

2. Secondary Outcome: Time to Mechanical Ventilation or Death up to Day 28
Description: Time to Mechanical Ventilation or Death defined as the time from randomization to the first occurrence of death or mechanical ventilation. For participants already on mechanical ventilation at baseline, only death is counted as an event.
Time Frame: Up to Day 28
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Remdesivir + Placebo (RDV+PBO) - mITT Population; Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population: The mITT population included all randomized participants who received any amount of TCZ or placebo (PBO), with participants grouped according to treatment assigned at randomization.
Arm/Group | Remdesivir + Placebo (RDV+PBO) - mITT Population | Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population
Number analyzed (Participants) | 210 | 430
Days | NA [NA to NA] — Value not estimable due to insufficient number of events | NA [NA to NA] — Value not estimable due to insufficient number of events
Statistical Analysis 1: Comparison: Remdesivir + Placebo (RDV+PBO) - mITT Population vs Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population; Test type: Superiority; p = 0.8993, Log Rank; Hazard Ratio (HR) = 0.980, 95% CI 2-sided [0.72 to 1.34]

3. Secondary Outcome: Clinical Status as Assessed by the Investigator Using a 7-category Ordinal Scale of Clinical Status on Day 14
Description: Clinical status was assessed by the investigator according to the following ordinal scale categories:
  1. Discharged (or "ready for discharge" as evidenced by normal temperature and respiratory rate, and stable oxygen saturation on ambient air or </= 2L supplemental oxygen)
  2. Non-intensive care unit (ICU) hospital ward (or "ready for hospital ward") not requiring supplemental oxygen
  3. Non-ICU hospital ward (or "ready for hospital ward") requiring supplemental oxygen
  4. ICU or non-ICU hospital ward, requiring non-invasive ventilation or high-flow oxygen
  5. ICU, requiring intubation and mechanical ventilation
  6. ICU, requiring extracorporeal membrane oxygenation (ECMO) or mechanical ventilation and additional organ support (e.g., vasopressors, renal replacement therapy)
  7. Death
Time Frame: Day 14
Population: Two participants in the RDV+TCZ arm had no post-baseline clinical status data to Day 14 and were excluded from analysis for this endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | Remdesivir + Placebo (RDV+PBO) - mITT Population | Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population
Number analyzed (Participants) | 210 | 428
Percentage of Participants
  Category 1 | 52.4 | 54.0
  Category 2 | 1.9 | 2.6
  Category 3 | 11.4 | 8.9
  Category 4 | 6.7 | 9.6
  Category 5 | 6.7 | 4.9
  Category 6 | 11.4 | 10.0
  Category 7 | 9.5 | 10.0
Statistical Analysis 1: Comparison: Remdesivir + Placebo (RDV+PBO) - mITT Population vs Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population; Test type: Superiority; p = 0.7648, Regression, Logistic; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.77 to 1.44]

4. Secondary Outcome: Time to Death up to Day 28
Description: Time to death is defined as the time from randomization to death.
Time Frame: Up to Day 28
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Remdesivir + Placebo (RDV+PBO) - mITT Population | Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population
Number analyzed (Participants) | 210 | 430
Days | NA [NA to NA] — Value not estimable due to insufficient number of events | NA [NA to NA] — Value not estimable due to insufficient number of events
Statistical Analysis 1: Comparison: Remdesivir + Placebo (RDV+PBO) - mITT Population vs Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population; Test type: Superiority; p = 0.7867, Log Rank; Hazard Ratio (HR) = 0.948, 95% CI 2-sided [0.65 to 1.39]

5. Secondary Outcome: Time to Death up to Day 60
Description: Time to death is defined as the time from randomization to death.
Time Frame: Up to Day 60
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Remdesivir + Placebo (RDV+Placebo) - mITT Population | Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population
Number analyzed (Participants) | 210 | 430
Days | NA [NA to NA] — Value not estimable due to insufficient number of events | NA [NA to NA] — Value not estimable due to insufficient number of events
Statistical Analysis 1: Comparison: Remdesivir + Placebo (RDV+Placebo) - mITT Population vs Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population; Test type: Superiority; p = 0.4602, Log Rank; Hazard Ratio (HR) = 0.882, 95% CI 2-sided [0.63 to 1.23]

6. Secondary Outcome: Time to Improvement of at Least 2 Categories Relative to Baseline on a 7-category Ordinal Scale of Clinical Status up to Day 28
Description: Defined as time from randomization to the time when at least a 2-category improvement in the 7-category ordinal scale is observed. Patients who die are censored at day 28.
  Clinical status was assessed by the investigator according to the following ordinal scale categories:
  1. Discharged (or "ready for discharge" as evidenced by normal temperature and respiratory rate, and stable oxygen saturation on ambient air or </= 2L supplemental oxygen)
  2. Non-intensive care unit (ICU) hospital ward (or "ready for hospital ward") not requiring supplemental oxygen
  3. Non-ICU hospital ward (or "ready for hospital ward") requiring supplemental oxygen
  4. ICU or non-ICU hospital ward, requiring non-invasive ventilation or high-flow oxygen
  5. ICU, requiring intubation and mechanical ventilation
  6. ICU, requiring extracorporeal membrane oxygenation (ECMO) or mechanical ventilation and additional organ support (e.g., vasopressors, renal replacement therapy)
  7. Death
Time Frame: Up to Day 28
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Remdesivir + Placebo (RDV+PBO) - mITT Population | Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population
Number analyzed (Participants) | 210 | 430
Days | 11.0 [10.0 to 13.0] | 12.0 [11.0 to 13.0]
Statistical Analysis 1: Comparison: Remdesivir + Placebo (RDV+PBO) - mITT Population vs Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population; Test type: Superiority; p = 0.8664, Log Rank; Hazard Ratio (HR) = 0.982, 95% CI 2-sided [0.80 to 1.21]

7. Secondary Outcome: Clinical Status as Assessed by the Investigator Using a 7-category Ordinal Scale of Clinical Status on Day 7
Description: as for outcome 3
Time Frame: Day 7
Population: Two participants in the RDV+TCZ arm had no post-baseline clinical status data to Day 7 and were excluded from analysis for this endpoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Remdesivir + Placebo (RDV+PBO) - mITT Population | Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population
Number analyzed (Participants) | 210 | 428
Percentage of participants
  Category 1 | 21.9 | 19.4
  Category 2 | 4.3 | 5.6
  Category 3 | 17.6 | 20.1
  Category 4 | 30.0 | 29.4
  Category 5 | 9.5 | 10.0
  Category 6 | 12.9 | 12.1
  Category 7 | 3.8 | 3.3
Statistical Analysis 1: Comparison: Remdesivir + Placebo (RDV+PBO) - mITT Population vs Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population; Test type: Superiority; p = 0.9569, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.75 to 1.35]

8. Secondary Outcome: Clinical Status as Assessed by the Investigator Using a 7-category Ordinal Scale of Clinical Status on Day 21
Description: as for outcome 3
Time Frame: Day 21
Population: Two participants in the RDV+TCZ arm had no post-baseline clinical status data to Day 21 and were excluded from analysis for this endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | Remdesivir + Placebo (RDV+PBO) - mITT Population | Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population
Number analyzed (Participants) | 210 | 428
Percentage of Participants
  Category 1 | 62.4 | 64.3
  Category 2 | 1.4 | 1.2
  Category 3 | 4.8 | 4.7
  Category 4 | 2.9 | 4.4
  Category 5 | 6.7 | 5.6
  Category 6 | 7.1 | 5.8
  Category 7 | 14.8 | 14.0
Statistical Analysis 1: Comparison: Remdesivir + Placebo (RDV+PBO) - mITT Population vs Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population; Test type: Superiority; p = 0.6331, Regression, Logistic; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.78 to 1.52]

9. Secondary Outcome: Clinical Status as Assessed by the Investigator Using a 7-category Ordinal Scale of Clinical Status on Day 28
Description: as for outcome 3
Time Frame: Day 28
Population: Two participants in the RDV+TCZ arm had no post-baseline clinical status data to Day 28 and were excluded from analysis for this endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | Remdesivir + Placebo (RDV+PBO) - mITT Population | Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population
Number analyzed (Participants) | 210 | 428
Percentage of Participants
  Category 1 | 67.1 | 66.4
  Category 2 | 1.4 | 1.4
  Category 3 | 1.0 | 3.5
  Category 4 | 2.9 | 3.0
  Category 5 | 4.3 | 3.7
  Category 6 | 3.8 | 3.7
  Category 7 | 19.5 | 18.2
Statistical Analysis 1: Comparison: Remdesivir + Placebo (RDV+PBO) - mITT Population vs Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population; Test type: Superiority; p = 0.9622, Regression, Logistic; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.70 to 1.40]

10. Secondary Outcome: Clinical Status as Assessed by the Investigator Using a 7-category Ordinal Scale of Clinical Status on Day 60
Description: as for outcome 3
Time Frame: Day 60
Population: Two participants in the RDV+TCZ arm had no post-baseline clinical status data to Day 60 and were excluded from analysis for this endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | Remdesivir + Placebo (RDV+PBO) - mITT Population | Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population
Number analyzed (Participants) | 210 | 428
Percentage of Participants
  Category 1 | 70.0 | 72.2
  Category 2 | 1.4 | 0.7
  Category 3 | 1.0 | 1.4
  Category 4 | 1.4 | 1.6
  Category 5 | 0.5 | 0.7
  Category 6 | 0 | 0.7
  Category 7 | 25.7 | 22.7
Statistical Analysis 1: Comparison: Remdesivir + Placebo (RDV+PBO) - mITT Population vs Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population; Test type: Superiority; p = 0.4850, Regression, Logistic; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.79 to 1.64]

11. Secondary Outcome: Proportion of Participants Requiring Initiation of Mechanical Ventilation Post-baseline (Participants Who Did Not Require Mechanical Ventilation at Baseline)
Description: Day 28: Participants who withdraw or die prior to Day 28 are assumed to have required mechanical ventilation. Participants without mechanical ventilation prior to discharge are assumed not to have required mechanical ventilation unless they die by Day 28, which are counted as an event.
  Day 60: Participants who withdraw or die prior to Day 60 are assumed to have required mechanical ventilation. Participants without mechanical ventilation prior to discharge are assumed not to have required mechanical ventilation unless they die by Day 60, which are counted as an event.
Time Frame: Day 28 and Day 60
Population: The analysis population for this endpoint included only participants not on mechanical ventilation at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Remdesivir + Placebo (RDV+PBO) - mITT Population | Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population
Number analyzed (Participants) | 188 | 371
Percentage of Participants
  Day 28 | 29.8 [23.3 to 36.3] | 27.5 [23.0 to 32.0]
  Day 60 | 31.4 [24.7 to 38.0] | 28.8 [24.2 to 33.5]
Statistical Analysis 1: Comparison: Remdesivir + Placebo (RDV+PBO) - mITT Population vs Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population; Day 28; Test type: Superiority; p = 0.5915, Cochran-Mantel-Haenszel; Weighted % difference = -2.2, 95% CI 2-sided [-10.2 to 5.9]
Statistical Analysis 2: Comparison: Remdesivir + Placebo (RDV+PBO) - mITT Population vs Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population; Day 60; Test type: Superiority; p = 0.5494, Cochran-Mantel-Haenszel; Weighted % difference = -2.5, 95% CI 2-sided [-10.5 to 5.6]

12. Secondary Outcome: Proportion of Participants Who Are Alive and Free of Respiratory Failure at Day 28 and Day 60 (Participants Requiring Mechanical Ventilation at Baseline)
Time Frame: Day 28 and Day 60
Population: The analysis population for this endpoint included only participants on mechanical ventilation at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Remdesivir + Placebo (RDV+PBO) - mITT Population | Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population
Number analyzed (Participants) | 22 | 59
Percentage of Participants
  Day 28 | 54.5 [33.7 to 75.4] | 40.7 [28.1 to 53.2]
  Day 60 | 63.6 [43.5 to 83.7] | 47.5 [34.7 to 60.2]
Statistical Analysis 1: Comparison: Remdesivir + Placebo (RDV+PBO) - mITT Population vs Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population; Day 28; Test type: Superiority; p = 0.2590, Cochran-Mantel-Haenszel; Weighted % difference = -14.1, 95% CI 2-sided [-37.4 to 9.2]
Statistical Analysis 2: Comparison: Remdesivir + Placebo (RDV+PBO) - mITT Population vs Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population; Day 60; Test type: Superiority; p = 0.2290, Cochran-Mantel-Haenszel; Weighted % difference = -14.6, 95% CI 2-sided [-37.0 to 7.8]

13. Secondary Outcome: Duration of Mechanical Ventilation (Participants Requiring Mechanical Ventilation at Baseline) up to Day 28
Description: Participants who die by Day 28 are assigned a duration of 28 days.
Time Frame: Up to Day 28
Population: The analysis population for this endpoint included only participants on mechanical ventilation at baseline.
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Remdesivir + Placebo (RDV+PBO) - mITT Population | Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population
Number analyzed (Participants) | 22 | 59
Days | 16.7 [11.9 to 21.5] | 19.6 [16.8 to 22.4]
Statistical Analysis 1: Comparison: Remdesivir + Placebo (RDV+PBO) - mITT Population vs Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population; Test type: Superiority; p = 0.2434, Regression, Linear; Mean Difference (Final Values) = 3.1125, 95% CI 2-sided [-2.16 to 8.38]

14. Secondary Outcome: Difference in Mortality at Days 14, 28, and 60
Time Frame: Days 14, 28, and 60
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Remdesivir + Placebo (RDV+PBO) - mITT Population | Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population
Number analyzed (Participants) | 210 | 430
Percentage of Participants
  Day 14 | 9.5 [5.6 to 13.5] | 10.0 [7.2 to 12.8]
  Day 28 | 19.5 [14.2 to 24.9] | 18.1 [14.5 to 21.8]
  Day 60 | 25.7 [19.8 to 31.6] | 22.6 [18.6 to 26.5]
Statistical Analysis 1: Comparison: Remdesivir + Placebo (RDV+PBO) - mITT Population vs Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population; Day 14; Test type: Superiority; p = 0.8222, Cochran-Mantel-Haenszel; Weighted % difference = 0.6, 95% CI 2-sided [-4.4 to 5.6]
Statistical Analysis 2: Comparison: Remdesivir + Placebo (RDV+PBO) - mITT Population vs Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population; Day 28; Test type: Superiority; p = 0.6944, Cochran-Mantel-Haenszel; Weighted % difference = -1.3, 95% CI 2-sided [-7.8 to 5.2]
Statistical Analysis 3: Comparison: Remdesivir + Placebo (RDV+PBO) - mITT Population vs Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population; Day 60; Test type: Superiority; p = 0.3919, Cochran-Mantel-Haenszel; Weighted % difference = -3.0, 95% CI 2-sided [-10.1 to 4.0]

15. Secondary Outcome: Time to Recovery up to Day 28
Description: Defined as the time from randomization to the time when an ordinal scale category of 2 (non-ICU hospital ward or "ready for hospital ward" not requiring supplemental oxygen) or better is observed, not followed by ordinal scale category >2 or death. Participants who die are censored at day 28.
  1. Discharged (or "ready for discharge" as evidenced by normal temperature and respiratory rate, and stable oxygen saturation on ambient air or </= 2L supplemental oxygen)
  2. Non-intensive care unit (ICU) hospital ward (or "ready for hospital ward") not requiring supplemental oxygen
  3. Non-ICU hospital ward (or "ready for hospital ward") requiring supplemental oxygen
  4. ICU or non-ICU hospital ward, requiring non-invasive ventilation or high-flow oxygen
  5. ICU, requiring intubation and mechanical ventilation
  6. ICU, requiring extracorporeal membrane oxygenation (ECMO) or mechanical ventilation and additional organ support (e.g., vasopressors, renal replacement therapy)
  7. Death
Time Frame: Up to Day 28
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Remdesivir + Placebo (RDV+PBO) - mITT Population | Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population
Number analyzed (Participants) | 210 | 430
Days | 13.0 [10.0 to 15.0] | 13.0 [11.0 to 14.0]
Statistical Analysis 1: Comparison: Remdesivir + Placebo (RDV+PBO) - mITT Population vs Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population; Test type: Superiority; p = 0.6778, Log Rank; Hazard Ratio (HR) = 0.957, 95% CI 2-sided [0.78 to 1.18]

16. Secondary Outcome: Proportion of Participants Who Are Discharged or "Ready for Discharge" up to Day 28
Description: Defined as hospital discharge or "Ready for Discharge" not followed by ordinal scale category >1, hospital readmission or death.
  1. Discharged (or "ready for discharge" as evidenced by normal temperature and respiratory rate, and stable oxygen saturation on ambient air or </= 2L supplemental oxygen)
  2. Non-intensive care unit (ICU) hospital ward (or "ready for hospital ward") not requiring supplemental oxygen
  3. Non-ICU hospital ward (or "ready for hospital ward") requiring supplemental oxygen
  4. ICU or non-ICU hospital ward, requiring non-invasive ventilation or high-flow oxygen
  5. ICU, requiring intubation and mechanical ventilation
  6. ICU, requiring extracorporeal membrane oxygenation (ECMO) or mechanical ventilation and additional organ support (e.g., vasopressors, renal replacement therapy)
  7. Death
Time Frame: Up to Day 28
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Remdesivir + Placebo (RDV+PBO) - mITT Population | Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population
Number analyzed (Participants) | 210 | 430
Percentage of participants | 67.1 [60.8 to 73.5] | 66.0 [61.6 to 70.5]
Statistical Analysis 1: Comparison: Remdesivir + Placebo (RDV+PBO) - mITT Population vs Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population; Test type: Superiority; p = 0.7692, Cochran-Mantel-Haenszel; Weighted % difference = -0.9, 95% CI 2-sided [-8.7 to 6.8]

17. Secondary Outcome: Proportion of Participants Who Require Initiation of Mechanical Ventilation Post-baseline or Die up to Day 28
Description: Participants already on mechanical ventilation at baseline are only counted as an event if death occurs.
Time Frame: Up to Day 28
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Remdesivir + Placebo (RDV+PBO) - mITT Population | Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population
Number analyzed (Participants) | 210 | 430
Percentage of participants | 29.0 [22.9 to 35.2] | 28.6 [24.3 to 32.9]
Statistical Analysis 1: Comparison: Remdesivir + Placebo (RDV+PBO) - mITT Population vs Remdesivir + Tocilizumab (RDV+TCZ) - mITT Population; Test type: Superiority; p = 0.9334, Cochran-Mantel-Haenszel; Weighted % difference = -0.3, 95% CI 2-sided [-7.8 to 7.2]

18. Other Pre Specified Outcome: Percentage of Participants With Adverse Events (AEs) Tabulated by Severity
Description: AEs were reported according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE).
  Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL) Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL Grade 4: Life-threatening consequences; urgent intervention indicated Grade 5: Death related to AE
  Participants are counted at the highest AE grade experienced.
Time Frame: Up to Day 60
Population: Participants that only received RDV and did not receive TCZ/PBO were included in the RDV+PBO arm of the safety population.
Measure: Number; unit: Percentage of participants
Groups:
- Remdesivir + Placebo (RDV+PBO) - Safety Population; Remdesivir + Tocilizumab (RDV+TCZ) - Safety Population: The safety population included all participants who received any amount of study medication (RDV and/or TCZ/PBO), with participants grouped according to the actual treatment received rather than the treatment assigned at randomization.
Arm/Group | Remdesivir + Placebo (RDV+PBO) - Safety Population | Remdesivir + Tocilizumab (RDV+TCZ) - Safety Population
Number analyzed (Participants) | 213 | 429
Percentage of participants
  Grade 1 | 9.9 | 10.5
  Grade 2 | 21.1 | 28.2
  Grade 3 | 10.3 | 11.2
  Grade 4 | 4.2 | 4.9
  Grade 5 | 25.8 | 22.6

19. Other Pre Specified Outcome: Proportion of Participants With Any Post-Treatment Infection
Time Frame: Up to Day 60
Population: as for outcome 18
Measure: Number; unit: Percentage of Participants
Arm/Group | Remdesivir + Placebo (RDV+PBO) - Safety Population | Remdesivir + Tocilizumab (RDV+TCZ) - Safety Population
Number analyzed (Participants) | 213 | 429
Percentage of Participants
  Serious infections | 27.7 | 22.6
  Infections | 35.7 | 33.3
  Opportunistic infections | 2.3 | 1.4

ADVERSE EVENTS:
Time Frame: Up to Day 60
Description: The safety analysis population consisted of all participants who received any amount of study medication (RDV and/or TCZ/PBO). Participants were grouped according to the treatment received rather than by the treatment assigned at randomization. Participants that only received RDV and did not receive TCZ/PBO were included in the RDV+PBO arm of the safety population.
Arm/Group | Remdesivir + Placebo (RDV+PBO) | Remdesivir + Tocilizumab (RDV+TCZ)
All-Cause Mortality (participants affected / at risk) | 55/213 | 97/429
Serious Adverse Events (participants affected / at risk) | 76/213 | 141/429
Other Adverse Events (participants affected / at risk) | 70/213 | 144/429
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remdesivir + Placebo (RDV+PBO) (N=213) | Remdesivir + Tocilizumab (RDV+TCZ) (N=429)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Bicytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 3 (3) | 2 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 3 (3)
Chronic left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Brain death (General disorders) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 1 (1) | 2 (3)
Death (General disorders) | 1 (1) | 2 (2)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 2 (2)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 2 (2)
Bacteraemia (Infections and infestations) | 2 (3) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 8 (8) | 14 (14)
COVID-19 pneumonia (Infections and infestations) | 27 (27) | 36 (36)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Fungaemia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6) | 21 (22)
Pneumonia acinetobacter (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 4 (4) | 5 (5)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 6 (7) | 11 (13)
Septic shock (Infections and infestations) | 10 (10) | 23 (23)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Systemic candida (Infections and infestations) | 2 (2) | 0 (0)
Tracheobronchitis (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 4 (4)
Urosepsis (Infections and infestations) | 2 (2) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1)
Brain herniation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood culture positive (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 3 (3) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Brain compression (Nervous system disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 5 (5)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 5 (5)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 2 (2) | 1 (1)
Haemorrhagic transformation stroke (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Neurotoxicity (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 14 (14) | 21 (21)
Renal failure (Renal and urinary disorders) | 0 (0) | 5 (5)
Renal impairment (Renal and urinary disorders) | 5 (5) | 1 (1)
Renal injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Aortic thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 1 (1)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 4 (4) | 4 (4)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 4 (4)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remdesivir + Placebo (RDV+PBO) (N=213) | Remdesivir + Tocilizumab (RDV+TCZ) (N=429)
Anaemia (Blood and lymphatic system disorders) | 14 (15) | 13 (13)
Constipation (Gastrointestinal disorders) | 25 (25) | 54 (54)
Urinary tract infection (Infections and infestations) | 11 (11) | 20 (21)
Transaminases increased (Investigations) | 10 (10) | 25 (25)
Hyperglycaemia (Metabolism and nutrition disorders) | 9 (9) | 22 (22)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (9) | 23 (26)
Acute kidney injury (Renal and urinary disorders) | 11 (11) | 24 (25)
Hypotension (Vascular disorders) | 12 (12) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT04409262/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT04409262/SAP_001.pdf